CLINICAL TRIAL: NCT00956007
Title: A Phase III Study of Postoperative Radiation Therapy (IMRT) +/- Cetuximab for Locally-Advanced Resected Head and Neck Cancer
Brief Title: RT With or Without Cetuximab in Treating Patients Who Have Undergone Surgery for Locally Advanced Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 0920; CDR0000651536; NCI-2011-00878 (Registry Identifier: CTRP (Clinical Trials Reporting Program); 5U10CA180868 (NIH); NCT01311063 (obsolete NCT alias)
Record Dates: First submitted 2009-08-08; First posted 2009-08-11 (Estimated); Results first posted 2024-05-28 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Cetuximab; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Intensity-Modulated Radiotherapy (Active Comparator): Radiation therapy: 60 Gy intensity-modulated radiotherapy (IMRT), 2 Gy/day in 30 fractions (5 days a week for 6 weeks).
  Interventions: Radiation: intensity-modulated radiation therapy
- Arm II: IMRT plus cetuximab (Experimental): Radiation therapy (RT): 60 Gy IMRT, 2 Gy/day in 30 fractions (5 days a week for 6 weeks).
  Cetuximab: 400 mg/m^2 intravenously (IV) at least 5 days prior to IMRT; 250 mg/m^2 IV once a week for 6 weeks during RT and continuing 4 weeks after RT.
  Interventions: Biological: cetuximab; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Biological: cetuximab — intravenously
  Arms: Arm II: IMRT plus cetuximab
Radiation: intensity-modulated radiation therapy — daily fractions

SUMMARY:
RATIONALE: Giving radiation therapy that uses a 3-dimensional (3-D) image of the tumor to help focus thin beams of radiation directly on the tumor, and giving radiation therapy in higher doses over a shorter period of time, may kill more tumor cells and have fewer side effects. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether radiation therapy is more effective when given alone or together with cetuximab in treating patients with head and neck cancer that has been removed by surgery.

PURPOSE: This randomized phase III trial is studying radiation therapy to see how well it works compared with radiation therapy given together with cetuximab in treating patients who have undergone surgery for locally advanced head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether the addition of cetuximab to postoperative intensity-modulated radiotherapy (IMRT) will improve overall survival (OS) in patients with locally advanced squamous cell carcinoma of the head and neck at intermediate risk following surgery.

Secondary

* Assess the impact of the addition of cetuximab to postoperative IMRT on disease-free survival (DFS) of these patients.
* Assess the impact of the addition of cetuximab to postoperative IMRT on acute and late dysphagia, xerostomia, skin toxicity, and other toxicities according to common Toxicity Criteria for Adverse Effects (CTCAE), v. 4 and their relationships with patient-reported outcomes at 3, 12, and 24 months.
* Analyze tumor for epidermal growth factor receptor (EGFR), specifically the extent of EGFR overexpression by immuno-histochemistry (IHC) and Fluorescence in situ hybridization (FISH) analysis, EGFRvIII expression, as well as the association of these assay data with OS and DFS.
* Analyze tumor for human papillomavirus (HPV) infection (as defined by in situ hybridization), specifically, within the cohort of patients with oropharynx cancer, to perform an exploratory analysis of the impact of HPV on DFS and OS of this patient subset.
* Analyze tumor DNA for TP53 mutations as a predictor of response to cetuximab and prognosis.
* Analyze germline DNA of polymorphic variants in EGFR intron repeats as a predictor of response to cetuximab.

Tertiary

* Assess the impact of the addition of cetuximab to postoperative IMRT on loco-regional control.
* Assess the impact of the addition of cetuximab to postoperative IMRT on patient-reported quality of life, swallowing, xerostomia, and skin toxicity based on head and neck specific instruments, including the Performance Status Scale for Head and Neck Cancer (PSS-HN), the Functional Assessment of Cancer Therapy-Head & Neck (FACT-H&N), the University of Michigan Xerostomia-Related Quality of Life Scale (XeQOLS), and the Dermatology Life Quality Index (DLQI).
* Assess the impact of the addition of cetuximab to postoperative IMRT on cost-utility analysis using the EuroQol (EQ-5D).
* Evaluate the utility of image-guided radiotherapy (IGRT) as a means of enhancing the efficacy (i.e., loco-regional control) of IMRT while reducing the acute and/or late toxicity (particularly xerostomia) and improving patient-reported outcomes (particularly XeQOLS scores).
* Retrospectively compare the loco-regional control rate in patients treated with IMRT alone (no IGRT or cetuximab) with similar patients treated with external beam radiotherapy alone in the postoperative clinical trial Radiation Therapy Oncology Group (RTOG)-95 01.

OUTLINE: This is a multicenter study. Patients are stratified according to clinical stage (T1-3 vs T4a), EGFR expression (high [≥ 80% of cells staining positive] vs low [< 80% of cells staining positive] vs not evaluable), primary site of disease (oral cavity vs larynx vs oropharynx p16+ vs oropharynx p16- vs oropharynx, p16 not evaluable), and use of image-guided radiotherapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo intensity-modulated radiotherapy (IMRT) once daily 5 days a week for 6 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo IMRT as in arm I. Patients also receive cetuximab IV over 1-2 hours once weekly beginning at least 5 days prior to the start of IMRT and continuing for 4 weeks after the completion of IMRT (for a total of 11 doses) in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and at 3, 12, and 24 months.

Tissue samples are collected periodically for further laboratory analysis.

After completion of study treatment, patients are followed up at 1 and 3 months, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Conditions for Patient Eligibility:

* Pathologically (histologically) proven diagnosis of squamous cell carcinoma (including variants such as verrucous carcinoma, spindle cell carcinoma, carcinoma NOS [not otherwise specified], etc.) of the head/neck (oral cavity, oropharynx or larynx); Note: Hypopharynx primaries are excluded because these patients have both a poor prognosis and high likelihood of post- radiation complications.
* Clinical stage T1, N1-2 or T2-4a, N0-2, M0 including no distant metastases, based upon the following minimum diagnostic workup:

  * General history and physical examination by a radiation oncologist and/or medical oncologist within 8 weeks prior to registration;
  * Examination by an otolaryngologists or Head & Neck Surgeon, within 8 weeks prior to registration; a laryngopharyngoscopy (mirror and/or fiberoptic and/or direct procedure) is recommended but not required.
  * Chest x-ray (at a minimum) or chest computed tomography (CT) scan (with or without contrast) or CT/positron emission tomography (PET) of chest (with or without contrast) within 8 weeks prior to registration.
* Gross total resection of the primary tumor with curative intent must be completed within 7 weeks of registration with surgical pathology demonstrating one or more of the following intermediate risk factors:

  * Perineural invasion;
  * Lymphovascular invasion;
  * Single lymph node > 3 cm or ≥ 2 lymph nodes (all < 6 cm) [no extracapsular extension];
  * Close margin(s) of resection, defined as cancer extending to within 5 mm of a surgical margin, and/or an initially focally positive margin that is subsequently superseded by intraoperative negative margins. Similarly, patients whose tumors had focally positive margins in the main specimen but negative margins from re-excised samples in the region of the positive margin are eligible.
  * Pathologically confirmed T3 or T4a primary tumor.
  * T2 oral cavity cancer with > 5 mm depth of invasion.
* Zubrod Performance Status of 0-1 within 2 weeks prior to registration;
* Age ≥ 18;
* Complete blood count (CBC)/differential obtained within 4 weeks prior to registration on study, with adequate bone marrow function defined as follows:

  * Absolute granulocyte count (AGC) ≥ 1,500 cells/mm3;
  * Platelets ≥ 100,000 cells/mm3;
  * Hemoglobin (Hgb) ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥8.0 g/dl is acceptable).
* Adequate hepatic function, defined as follows:

  * Total bilirubin < 2 x institutional upper limit of normal (ULN) within 2 weeks prior to registration;
  * aspartate aminotransferase (AST) or alanine transaminase (ALT) < 3 x institutional ULN within 2 weeks prior to registration.
* Adequate renal function, defined as follows:

  * Serum creatinine (Scr) < 2 x institutional ULN within 2 weeks prior to registration or; creatinine clearance (CCr) ≥ 50 ml/min within 2 weeks prior to registration determined by 24-hour collection or estimated by Cockcroft-Gault formula: CCr male = [(140 - age) x (weight in kg)] /[(SCr mg/dl) x (72)] CCr female = 0.85 x (CCr male)
* Negative serum pregnancy test within 2 weeks prior to registration for women of childbearing potential;
* The following assessments are required within 2 weeks prior to the start of registration:

Na, K, Cl, glucose, Ca, Mg, and albumin. Note: Patients with an initial magnesium < 0.5 mmol/L (1.2 mg/dl) may receive corrective magnesium supplementation but should continue to receive either prophylactic weekly infusion of magnesium and/or oral magnesium supplementation (e.g., magnesium oxide) at the investigator's discretion.

* Women of childbearing potential and male participants who are sexually active must agree to use a medically effective means of birth control;
* Patients must provide study specific informed consent prior to study entry, including consent for mandatory tissue submission for EGFR and for oropharyngeal patients, HPV analyses.

Conditions for Patient Ineligibility

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years; noninvasive cancers (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible) are permitted even if diagnosed and treated < 3 years ago. Patients with simultaneous primaries or bilateral tumors are excluded, with the exception of patients with bilateral tonsil cancers or patients with T1-2, N0, M0 resected differentiated thyroid carcinoma, who are eligible.
* Per the operative and/or pathology report, positive margin(s) [defined as tumor present at the cut or inked edge of the tumor], nodal extracapsular extension, and/or gross residual disease after surgery; Note: Patients whose tumors had focally positive margins in the main specimen but negative margins from re-excised samples in the region of the positive margin are eligible.
* Prior systemic chemotherapy or anti-EGF therapy for the study cancer; note: prior chemotherapy or anti-EGF therapy for a different cancer is allowable.
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields;
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within 6 months prior to registration;
  * Transmural myocardial infarction within 6 months prior to registration;
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration;
  * Idiopathic pulmonary fibrosis or other severe interstitial lung disease that requires oxygen therapy or is thought to require oxygen therapy within 1 year prior to registration;
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for coagulation parameters are not required for entry into this protocol.
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note: HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
  * Grade 3-4 electrolyte abnormalities (CTCAE v4):
* Serum calcium (ionized or adjusted for albumin) < 7 mg/dl (1.75 mmol/L) or >12.5 mg/dl (> 3.1 mmol/L) despite intervention to normalize levels;
* Glucose < 40 mg/dl (< 2.2 mmol/L) or > 250 mg/dl (> 14mmol/L);
* Magnesium < 0.9 mg/dl (< 0.4 mmol/L) or > 3 mg/dl (> 1.23 mmol/L) despite intervention to normalize levels;
* Potassium < 3.0 mmol/L or > 6 mmol/L despite intervention to normalize levels;
* Sodium < 130 mmol/L or > 155 mmol/L despite intervention to normalize levels.
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
* Prior allergic reaction to cetuximab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2010-03-31 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2029-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Machtay, MD, Study Chair — Milton S. Hershey Medical Center, Penn State Health
Locations (264):
- United States (250):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Oncology Associates-West Orange Grove, Tucson, Arizona
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - City of Hope, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - University of Southern California/Norris Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Bay Area Tumor Institute CCOP, Oakland, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - University of California at Davis Cancer Center, Sacramento, California
  - Mercy General Hospital Radiation Oncology Center, Sacramento, California
  - UCSF-Mount Zion, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Saint Helena Hospital, St. Helena, California
  - Stanford University Hospitals and Clinics, Stanford, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Yale University, New Haven, Connecticut
  - William Backus Hospital, Norwich, Connecticut
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - University of Miami Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Joseph's-Candler Health System, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Hines Veterans Administration Hospital, Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Community Regional Cancer Care-East Radiation Oncology, Indianapolis, Indiana
  - Community Regional Cancer Care-North, Indianapolis, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Touro Infirmary, New Orleans, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Cape Radiation Oncology, Cape Girardeau, Missouri
  - Siteman Cancer Center - Saint Peters, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Kansas City Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - The Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Exeter Hospital, Exeter, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - UMDNJ - New Jersey Medical School, Newark, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - New York Oncology Hematology PC - Albany, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Sands Cancer Center, Canandaigua, New York
  - Memorial Sloan Kettering Cancer Center Commack, Commack, New York
  - Beth Israel Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University Radiation Oncology, Rochester, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan-Kettering Cancer Center Rockville Centre, Rockville Centre, New York
  - Memorial Sloan-Kettering Cancer Center at Sleepy Hallow, Sleepy Hollow, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Cancer Centers of North Carolina, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Geaugra Hospital, Chardon, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Summa Health Center at Lake Medina, Medina, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center Ireland Cancer Center, Middleburg Heights, Ohio
  - UHHS-Chagrin Highlands Medical Center, Orange, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Robinson Radiation Oncology, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Cancer Center-Strongsville, Strongsville, Ohio
  - Flower Hospital, Sylvania, Ohio
  - University Pointe, West Chester, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Specialty Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Western Oncology Research Consortium, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Portland Veterans Administration Medical Center, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Health System Cancer Institute/Greenville CCOP, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology PA - Bedford, Bedford, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Oncology-Denton South, Denton, Texas
  - The Klabzuba Cancer Center, Fort Worth, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Texas Oncology-Seton Williamson, Round Rock, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - Cancer Care Centers of South Texas- Northeast, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Cancer Center-Sherman, Sherman, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Texas Oncology-Wichita Falls Texoma Cancer Center, Wichita Falls, Texas
  - Intermountain Medical Center, Murray, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - University of Virginia, Charlottesville, Virginia
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Sentara Hospitals, Norfolk, Virginia
  - Hunter Holmes McGuire Veterans Administration Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - Harrison Medical Center, Bremerton, Washington
  - Tri-Cities Cancer Center, Kennewick, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - Northwest CCOP, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology, Appleton, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Clement J. Zablocki VA Medical Center, Milwaukee, Wisconsin
  - Door County Cancer Center, Sturgeon Bay, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
- Canada (12):
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Health Sciences North, Greater Sudbury, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute-General Division, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - CHUQ - Pavilion Hotel-Dieu de Quebec, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Chinese University of Hong Kong-Prince of Wales Hospital, Shatin, Hong Kong, China
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Machtay M, Torres-Saavedra PA, Thorstad W, Nguyen-Tan PF, Siu LL, Holsinger FC, El-Naggar A, Chung C, Cmelak A, Burtness B, Bednarz G, Quon H, Breen SL, Gwede CK, Dicker AP, Yao M, Jordan RC, Dorth J, Lee N, Chan JW, Dunlap N, Bar-Ad V, Stokes WA, Chakravarti A, Sher D, Rao S, Harris J, Yom SS, Le QT; NRG Oncology RTOG 0920 Collaborating Team. Postoperative Radiotherapy +/- Cetuximab for Intermediate-Risk Head and Neck Cancer. J Clin Oncol. 2025 Apr 20;43(12):1474-1487. doi: 10.1200/JCO-24-01829. Epub 2025 Jan 22. PMID 39841939

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After trial registration, tissue slides from the tumor specimen were sent to the NRG Oncology biorepository for immunohistochemical analysis of epidermal growth factor receptor (EGFR) expression and (for oropharynx cancer) p16, a surrogate biomarker for human papillomavirus (HPV) positivity. From 702 registered participants, 627 were randomized.
Groups:
- IMRT: Radiation therapy: 60 Gy intensity-modulated radiotherapy (IMRT), 2 Gy/day in 30 fractions (5 days a week for 6 weeks).
- IMRT Plus Cetuximab: Radiation therapy (RT): 60 Gy IMRT, 2 Gy/day in 30 fractions (5 days a week for 6 weeks).
  Cetuximab: 400 mg/m^2 intravenously (IV) at least 5 days prior to IMRT; 250 mg/m^2 IV once a week for 6 weeks during RT and continuing 4 weeks after RT.
Period: Overall Study
Arm/Group | IMRT | IMRT Plus Cetuximab
Started | 314 | 313
Eligible | 287 | 290
Eligible and Started Protocol Treatment (Adverse event population) | 282 | 276
Completed (Participants contributing data to results are considered to have completed the study.) | 287 | 290
Not Completed | 27 | 23
Not completed — Protocol Violation | 27 | 23

BASELINE CHARACTERISTICS:
Population: Randomized eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | IMRT | IMRT Plus Cetuximab | Total
Number analyzed (Participants) | 287 | 290 | 577
Age, Continuous [Median (Full Range); unit: years] | 57 [27 to 80] | 57.5 [20 to 79] | 57 [20 to 80]
Age, Customized [Count of Participants; unit: Participants]
  ≤ 49 years | 62 | 71 | 133
  50 - 59 years | 111 | 95 | 206
  60 - 69 years | 91 | 101 | 192
  ≥ 70 years | 23 | 23 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 90 | 173
  Male | 204 | 200 | 404
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 16 | 38
  Not Hispanic or Latino | 256 | 268 | 524
  Unknown or Not Reported | 9 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 8 | 12 | 20
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 21 | 21 | 42
  White | 249 | 249 | 498
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 6 | 6 | 12
Zubrod performance status [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death
  Participants
    0 | 134 | 152 | 286
    1 | 153 | 138 | 291
Smoking history [Count of Participants; unit: Participants]
  Never | 92 | 110 | 202
  Former | 173 | 160 | 333
  Current | 21 | 18 | 39
  Unknown | 1 | 2 | 3
Smoking history: pack-years [Count of Participants; unit: Participants] — Population: Randomized eligible participants with data
  Participants
    number analyzed (Participants) | 251 | 259 | 510
    ≤ 10 | 139 | 152 | 291
    > 10 | 112 | 107 | 219
Type of radiation therapy [Count of Participants; unit: Participants]
  Intensity-modulated radiation therapy (IMRT) | 129 | 146 | 275
  IMRT+ image-guided radiation therapy (IGRT) | 153 | 128 | 281
  None | 5 | 16 | 21
EGFR expression [Count of Participants; unit: Participants]
  High (≥ 80% of cells positive) | 246 | 242 | 488
  Low (< 80% of cells positive) | 38 | 44 | 82
  Not evaluable | 3 | 4 | 7
Primary site [Count of Participants; unit: Participants]
  Oral cavity | 183 | 184 | 367
  Larynx | 44 | 38 | 82
  Oropharynx, p16-positive | 50 | 55 | 105
  Oropharynx, p16-negative | 6 | 8 | 14
  Oropharynx, p16 unknown | 4 | 5 | 9
Pathologic T stage [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 6th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    T1 | 54 | 55 | 109
    T2 | 120 | 116 | 236
    T3 | 42 | 51 | 93
    T4a | 71 | 68 | 139
Pathologic N stage [Count of Participants; unit: Participants] — Regional lymph nodes staging per AJCC 6th ed. refers to the number and/or extent of spread of lymph nodes that contain cancer. N0 means lymph nodes aren't involved. A higher number means the cancer is in more lymph nodes, farther away from the original tumor. NX means the lymph nodes cannot be assessed.
  Participants
    N0 | 101 | 105 | 206
    N1 | 56 | 62 | 118
    N2a | 15 | 13 | 28
    N2b | 88 | 99 | 187
    N2c | 23 | 6 | 29
    NX | 4 | 5 | 9
Pathologic AJCC stage [Count of Participants; unit: Participants] — Overall cancer stage per American Joint Committee on Cancer (AJCC) 6th ed. combines tumor (T), regional lymph node (N), and distant metastasis (M) staging to determine an overall stage of 0, I, II, III, or IV, ranging from least to most advanced, respectively. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. The higher the number after the N, the greater the involvement of regional lymph nodes. M0 indicates no distant metastasis.
  Participants
    Stage I (T1, N0, M0) | 7 | 6 | 13
    Stage II (T2, N0, M0) | 33 | 38 | 71
    Stage III (T3, N0, M0; T1-3, N1, M0) | 63 | 71 | 134
    Stage IV (T4a, N0-2, M0; any T, N2, M0; T4b, any N, M0; any T, N3, M0; any T, Any N, M1) | 182 | 171 | 353
    Unknown | 2 | 4 | 6
Number of intermediate risk factors (centrally reviewed) [Count of Participants; unit: Participants] — The following are considered "intermediate" risk factors:
  * Perineural invasion;
  * Lymphovascular invasion;
  * Single lymph node > 3 cm or ≥2 lymph nodes (all < 6 cm) [no extracapsular extension];
  * Close margin(s) of resection (close margins defined as cancer extending to within 5 mm of a surgical margin);
  * T3 or T4a primary tumor;
  * T2 oral cavity cancer with > 5 mm depth of invasion.
  Participants
    1 | 36 | 46 | 82
    2 | 121 | 105 | 226
    3 | 92 | 92 | 184
    4 | 30 | 37 | 67
    5 | 8 | 9 | 17
    6 | 0 | 1 | 1
Perineural invasion (centrally reviewed) [Count of Participants; unit: Participants]
  No | 161 | 148 | 309
  Yes | 114 | 121 | 235
  Indeterminate | 2 | 0 | 2
  Unknown | 10 | 21 | 31
Lymphovascular invasion (centrally reviewed) [Count of Participants; unit: Participants]
  No | 196 | 179 | 375
  Yes | 73 | 83 | 156
  Indeterminate | 5 | 5 | 10
  Unknown | 13 | 23 | 36
Lymph node > 3cm or multiple lymph nodes (centrally reviewed) [Count of Participants; unit: Participants]
  No | 160 | 155 | 315
  Yes | 119 | 121 | 240
  Indeterminate | 2 | 0 | 2
  Unknown | 6 | 14 | 20
Close margins of resection (centrally reviewed) [Count of Participants; unit: Participants] — "Close margin(s) of resection" is defined as cancer extending to within 5 mm of a surgical margin, and/or an initially focally positive margin that is subsequently superseded by intraoperative negative margins.
  Participants
    No | 39 | 33 | 72
    Yes | 226 | 223 | 449
    Indeterminate | 1 | 4 | 5
    Unknown | 21 | 30 | 51
T3 or microscopic T4a (centrally reviewed) [Count of Participants; unit: Participants]
  No | 175 | 179 | 354
  Yes | 110 | 109 | 219
  Unknown | 2 | 2 | 4
T2 oral cavity with >5mm depth of invasion (centrally reviewed) [Count of Participants; unit: Participants]
  No | 203 | 207 | 410
  Yes | 72 | 74 | 146
  Unknown | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Alive (Overall Survival)
Description: Overall survival time is defined as time from registration/randomization to the date of death from any cause or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method. Analysis occurred after all participants had potentially been on study for at least 5 years. The distributions of survival times are compared, which is reported in the statistical analysis results. Five-year rates are provided.
Time Frame: From randomization to date of death or last follow-up. Maximum follow-up at time of analysis was 12.1 years.
Population: Randomized eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT | IMRT Plus Cetuximab
Number analyzed (Participants) | 287 | 290
percentage of participants | 68.7 [63.1 to 74.3] | 76.5 [71.4 to 81.6]
Statistical Analysis 1: Comparison: IMRT vs IMRT Plus Cetuximab; This trial was designed to detect a hazard ratio (HR) of 0.74 with 80% statistical power and overall one-sided alpha of 0.025 (372 deaths) using a stratified log-rank test, assuming a control arm 3-year survival rate of 60.1%. The amended protocol based on ≥ 5 years potential follow-up projected 169 events, providing 55%, 66%, and 79% power to detect HRs of 0.71, 0.68, and 0.64, respectively, using the original one-sided alpha of 0.0183 the final analysis; Test type: Superiority; p = 0.0747, Log Rank — One-sided significance level = 0.0183; Stratified by EGFR and site/p16 status; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.60 to 1.08] — Stratified by EGFR and site/p16 status. Reference level = IMRT

2. Secondary Outcome: Percentage of Participants With ≥ Grade 3 Acute Dysphagia, Dry Mouth, or Skin Toxicity Related to Protocol Treatment
Description: Common Terminology Criteria for Adverse Events (version 4.0) grades adverse event severity from 1=mild to 5=death. Adverse events (AEs) assessed to be definitely, probably, or possibly related to protocol treatment were included. If relationship was missing, it was assumed to be definitely, probably, or possibly related to protocol treatment. Acute adverse events are those occurring within 90 days of the start of radiation therapy.
Time Frame: From start of radiation therapy to 90 days
Population: Randomized eligible participants who started protocol treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT | IMRT Plus Cetuximab
Number analyzed (Participants) | 282 | 276
percentage of participants
  Dysphagia | 13.1 [9.7 to 17.6] | 21.7 [17.3 to 27.0]
  Dry mouth (xerostomia) | 3.5 [1.9 to 6.4] | 1.8 [0.8 to 4.2]
  Dermatitis radiation | 6.4 [4.1 to 9.9] | 17.0 [13.1 to 21.9]
  Rash acneiform | 0.0 [0.0 to 1.3] | 13.4 [9.9 to 17.9]
Statistical Analysis 1: Comparison: IMRT vs IMRT Plus Cetuximab; Dysphagia; Test type: Superiority; p = 0.0075, Fisher Exact
Statistical Analysis 2: Comparison: IMRT vs IMRT Plus Cetuximab; Dry mouth; Test type: Superiority; p = 0.2955, Fisher Exact
Statistical Analysis 3: Comparison: IMRT vs IMRT Plus Cetuximab; Dermatitis radiation; Test type: Superiority; p = 0.0001, Fisher Exact
Statistical Analysis 4: Comparison: IMRT vs IMRT Plus Cetuximab; Rach acneiform; Test type: Superiority; p < 0.0001, Fisher Exact

3. Secondary Outcome: Percentage of Participants With Other ≥ Grade 3 Adverse Events Related to Protocol Treatment
Description: Adverse events other than dysphagia, dermatitis radiation, and rash acneiform. Common Terminology Criteria for Adverse Events (version 4.0) grades adverse event severity from 1=mild to 5=death. Adverse events (AEs) assessed to be definitely, probably, or possibly related to protocol treatment were included. If relationship was missing, it was assumed to be definitely, probably, or possibly related to protocol treatment. Acute adverse events are those occurring within 90 days of the start of radiation therapy.
Time Frame: From start of radiation therapy to 90 days.
Population: Randomized eligible participants who started protocol treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT | IMRT Plus Cetuximab
Number analyzed (Participants) | 282 | 276
percentage of participants | 33.0 [27.8 to 38.7] | 64.1 [58.3 to 69.6]
Statistical Analysis 1: Comparison: IMRT vs IMRT Plus Cetuximab; Test type: Superiority; p < 0.0001, Fisher Exact

4. Secondary Outcome: Percentage of Participants With ≥ Grade 3 Late Dysphagia, Dry Mouth, or Skin Toxicity Related to Protocol Treatment
Description: Common Terminology Criteria for Adverse Events (version 4.0) grades adverse event severity from 1=mild to 5=death. Adverse events assessed to be definitely, probably, or possibly related to protocol treatment were included. If relationship was missing, it was assumed to be definitely, probably, or possibly related to protocol treatment. Late adverse events are those occurring after days from the start of radiation therapy.
Time Frame: From 91 days after start of radiation therapy to date of last reported follow-up. Maximum follow-up at time of analysis was 12.1 years.
Population: Randomized eligible participants who started protocol treatment and had follow-up data at or after day 91 from start of radiation therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT | IMRT Plus Cetuximab
Number analyzed (Participants) | 279 | 268
percentage of participants
  Dysphagia | 8.6 [5.8 to 12.5] | 12.3 [8.9 to 16.8]
  Dry mouth (xerostomia) | 3.2 [1.7 to 6.0] | 1.5 [0.6 to 3.8]
  Dermatitis radiation | 1.4 [0.6 to 3.6] | 2.2 [1.0 to 4.8]
  Rash acneiform | 0.0 [0.0 to 1.4] | 1.5 [0.6 to 3.8]
Statistical Analysis 1: Comparison: IMRT vs IMRT Plus Cetuximab; Dysphagia; Test type: Superiority; p = 0.1641, Fisher Exact
Statistical Analysis 2: Comparison: IMRT vs IMRT Plus Cetuximab; Dry mouth; Test type: Superiority; p = 0.2623, Fisher Exact
Statistical Analysis 3: Comparison: IMRT vs IMRT Plus Cetuximab; Dermatitis radiation; Test type: Superiority; p = 0.5378, Fisher Exact
Statistical Analysis 4: Comparison: IMRT vs IMRT Plus Cetuximab; Rash acneiform; Test type: Superiority; p = 0.0570, Fisher Exact

5. Secondary Outcome: Percentage of Participants With Other ≥ Grade 3 Late Adverse Events Related to Protocol Treatment
Description: Adverse events other than dysphagia, dermatitis radiation, and rash acneiform. Common Terminology Criteria for Adverse Events (version 4.0) grades adverse event severity from 1=mild to 5=death. Adverse events (AEs) assessed to be definitely, probably, or possibly related to protocol treatment were included. If relationship was missing, it was assumed to be definitely, probably, or possibly related to protocol treatment. Late adverse events are those occurring after days from the start of radiation therapy.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT | IMRT Plus Cetuximab
Number analyzed (Participants) | 279 | 268
percentage of participants | 20.8 [16.4 to 25.9] | 26.1 [21.2 to 31.7]
Statistical Analysis 1: Comparison: IMRT vs IMRT Plus Cetuximab; Test type: Superiority; p = 0.1575, Fisher Exact

6. Secondary Outcome: Disease-free Survival
Description: Disease is defined as local-regional progression/recurrence (LRR) or distant metastasis (DM). LRR is defined as recurrent cancer in the tumor bed and/or neck not clearly attributable to a second primary neoplasm; both imaging and biopsy confirmation are strongly recommended. DM is defined as clear evidence of distant metastases; biopsy is recommended where possible. Disease-free survival time is defined as time from randomization to the date of first disease, death, or last known follow-up (censored), whichever occurred first. Disease-free survival rates are estimated using the Kaplan-Meier method. Analysis occurred after all participants had potentially been on study for at least 5 years. The distributions of disease-free survival times are compared, which is reported in the statistical analysis results. Five-year rates are provided.
Time Frame: From randomization to date of LRR, DM, death or last known follow-up, whichever occurred first. Maximum follow-up at time of analysis was 12.1 years.
Population: Randomized eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT | IMRT Plus Cetuximab
Number analyzed (Participants) | 287 | 290
percentage of participants | 63.6 [57.8 to 69.3] | 71.7 [66.3 to 77.1]
Statistical Analysis 1: Comparison: IMRT vs IMRT Plus Cetuximab; Test type: Superiority; p = 0.0168, Log Rank — One-sided; Stratified by EGFR and site/p16 status; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.57 to 0.98] — Stratified by EGFR and site/p16 status. Reference level = IMRT

7. Other Pre Specified Outcome: Xerostomia as Measured by University of Michigan Xerostomia-Related Quality of Life Scale (XeQOLS) at Baseline and at 3, 12, and 24 Months
Time Frame: From randomization to 2 years.
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Swallowing as Measured by the Normalcy of Diet Subscale of the Performance Status Scale for Head and Neck Cancer (PSS-HN) at Baseline and at 3, 12, and 24 Months
Time Frame: From randomization to 2 years.
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Skin Toxicity as Measured by the Dermatology Life Quality Index (DLQI) at Baseline and at 3, 12, and 24 Months
Time Frame: From randomization to 2 years.
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Quality of Life as Measured by Functional Assessment of Cancer Therapy-Head & Neck (FACT-HN) and EuroQol (EQ-5D) at Baseline and at 3, 12, and 24 Months
Time Frame: From randomization to 2 years.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Loco-regional Control
Time Frame: From randomization to date of failure (local or regional progression or distant progression or death) or last follow-up. Analysis occurs at the same time as the primary outcome.
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Percentage of Participants Alive (Overall Survival) by Sex
Description: as for outcome 1
Time Frame: From randomization to date of death or last follow-up. Maximum follow-up at time of analysis was 12.1 years.
Population: Randomized eligible participants. Data were stratified by sex.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT | IMRT Plus Cetuximab
Number analyzed (Participants) | 287 | 290
percentage of participants
  Female: number analyzed (Participants) | 83 | 90
  Female | 75.3 [65.8 to 84.7] | 72.1 [62.4 to 81.8]
  Male: number analyzed (Participants) | 204 | 200
  Male | 65.9 [59.0 to 72.7] | 78.5 [72.6 to 84.4]

13. Other Pre Specified Outcome: Percentage of Participants Alive (Overall Survival) by Ethnicity
Description: NIH-required analysis. Overall survival time is defined as time from registration/randomization to the date of death from any cause or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method. Analysis occurred after all participants had potentially been on study for at least 5 years. The distributions of survival times are compared, which is reported in the statistical analysis results. Five-year rates are provided.
Time Frame: From randomization to date of death or last follow-up. Maximum follow-up at time of analysis was 12.1 years.
Population: Randomized eligible participants. Data were stratified by ethnicity.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT | IMRT Plus Cetuximab
Number analyzed (Participants) | 287 | 290
percentage of participants
  Hispanic or Latino: number analyzed (Participants) | 22 | 16
  Hispanic or Latino | 81.8 [65.7 to 97.9] | 80.0 [59.8 to 100]
  Not Hispanic or Latino: number analyzed (Participants) | 256 | 268
  Not Hispanic or Latino | 66.9 [60.9 to 72.9] | 76.2 [70.9 to 81.5]
  Unknown or Not Reported: number analyzed (Participants) | 9 | 6
  Unknown or Not Reported | 88.9 [68.4 to 100] | 83.3 [53.5 to 100]

14. Other Pre Specified Outcome: Percentage of Participants Alive (Overall Survival) by Race
Description: as for outcome 13
Time Frame: From randomization to date of death or last follow-up. Maximum follow-up at time of analysis was 12.1 years.
Population: Randomized eligible participants. Data were stratified by race.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT | IMRT Plus Cetuximab
Number analyzed (Participants) | 287 | 290
percentage of participants
  American Indian or Alaska Native: number analyzed (Participants) | 0 | 2
  American Indian or Alaska Native |  | 0 [NA to NA] — Cannot be calculated because the participant was censored prior to the timepoint.
  Asian: number analyzed (Participants) | 8 | 12
  Asian | 53.6 [14.2 to 92.9] | 91.7 [76.0 to 100]
  Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 1 | 0
  Native Hawaiian or Other Pacific Islander | 0 [NA to NA] — Cannot be calculated because the participant was censored prior to the timepoint. |
  Black or African American: number analyzed (Participants) | 21 | 21
  Black or African American | 57.9 [35.7 to 80.1] | 69.6 [49.3 to 90.0]
  White: number analyzed (Participants) | 249 | 249
  White | 70.1 [64.2 to 76.0] | 76.8 [71.3 to 82.3]
  More than one race: number analyzed (Participants) | 2 | 0
  More than one race | 50.0 [0 to 100] |
  Unknown for Not Reported: number analyzed (Participants) | 6 | 6
  Unknown for Not Reported | 83.3 [53.5 to 100] | 80.0 [44.9 to 100]

ADVERSE EVENTS:
Time Frame: From randomization to date of death or last follow-up. Maximum follow-up at time of analysis was 12.1 years.
Description: All-cause mortality was assessed in randomized eligible participants. Adverse events were assessed in randomized eligible participants who started protocol treatment.
Arm/Group | IMRT | IMRT Plus Cetuximab
All-Cause Mortality (participants affected / at risk) | 97/287 | 87/290
Serious Adverse Events (participants affected / at risk) | 50/282 | 83/276
Other Adverse Events (participants affected / at risk) | 278/282 | 275/276
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT (N=282) | IMRT Plus Cetuximab (N=276)
Anemia (Blood and lymphatic system disorders) | 3 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Heart failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Eye disorders - Other (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 5 | 2
Duodenal hemorrhage (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 7 | 12
Esophageal fistula (Gastrointestinal disorders) | 0 | 1
Esophageal pain (Gastrointestinal disorders) | 1 | 0
Esophageal stenosis (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 8 | 18
Nausea (Gastrointestinal disorders) | 2 | 6
Oral pain (Gastrointestinal disorders) | 5 | 4
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 8
Chills (General disorders) | 0 | 1
Edema limbs (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 1
Fever (General disorders) | 1 | 5
Infusion related reaction (General disorders) | 0 | 4
Malaise (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 1
Anaphylaxis (Immune system disorders) | 0 | 2
Catheter related infection (Infections and infestations) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 1 | 3
Infective myositis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 2 | 3
Mucosal infection (Infections and infestations) | 0 | 2
Paronychia (Infections and infestations) | 0 | 1
Salivary gland infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 2
Skin infection (Infections and infestations) | 2 | 2
Soft tissue infection (Infections and infestations) | 1 | 1
Stoma site infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 4 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 | 3
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 3 | 3
Lymphocyte count increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Weight loss (Investigations) | 2 | 0
White blood cell decreased (Investigations) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 6 | 12
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 4 | 3
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 1
Aphonia (Nervous system disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Myelitis (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 2
Stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 2 | 0
Hallucinations (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 2
Hypotension (Vascular disorders) | 2 | 3
Thromboembolic event (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT (N=282) | IMRT Plus Cetuximab (N=276)
Anemia (Blood and lymphatic system disorders) | 39 | 74
Ear pain (Ear and labyrinth disorders) | 17 | 23
Hearing impaired (Ear and labyrinth disorders) | 33 | 40
Hyperthyroidism (Endocrine disorders) | 3 | 16
Hypothyroidism (Endocrine disorders) | 43 | 53
Abdominal pain (Gastrointestinal disorders) | 6 | 21
Constipation (Gastrointestinal disorders) | 39 | 80
Diarrhea (Gastrointestinal disorders) | 20 | 40
Dry mouth (Gastrointestinal disorders) | 253 | 246
Dyspepsia (Gastrointestinal disorders) | 13 | 24
Dysphagia (Gastrointestinal disorders) | 244 | 250
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 50 | 57
Mucositis oral (Gastrointestinal disorders) | 224 | 232
Nausea (Gastrointestinal disorders) | 83 | 121
Oral pain (Gastrointestinal disorders) | 105 | 114
Salivary duct inflammation (Gastrointestinal disorders) | 18 | 21
Vomiting (Gastrointestinal disorders) | 45 | 63
Chills (General disorders) | 6 | 18
Edema face (General disorders) | 21 | 23
Edema limbs (General disorders) | 5 | 16
Facial pain (General disorders) | 16 | 13
Fatigue (General disorders) | 165 | 192
Fever (General disorders) | 6 | 19
General disorders and administration site conditions - Other (General disorders) | 10 | 16
Localized edema (General disorders) | 18 | 9
Neck edema (General disorders) | 33 | 19
Pain (General disorders) | 68 | 66
Infections and infestations - Other (Infections and infestations) | 11 | 23
Mucosal infection (Infections and infestations) | 24 | 28
Dermatitis radiation (Injury, poisoning and procedural complications) | 223 | 212
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 13 | 20
Alanine aminotransferase increased (Investigations) | 10 | 34
Alkaline phosphatase increased (Investigations) | 12 | 19
Aspartate aminotransferase increased (Investigations) | 15 | 28
Lymphocyte count decreased (Investigations) | 48 | 87
Platelet count decreased (Investigations) | 10 | 15
Weight loss (Investigations) | 106 | 126
White blood cell decreased (Investigations) | 22 | 38
Anorexia (Metabolism and nutrition disorders) | 76 | 92
Dehydration (Metabolism and nutrition disorders) | 23 | 28
Hypercalcemia (Metabolism and nutrition disorders) | 7 | 15
Hyperglycemia (Metabolism and nutrition disorders) | 21 | 44
Hyperkalemia (Metabolism and nutrition disorders) | 7 | 19
Hypoalbuminemia (Metabolism and nutrition disorders) | 13 | 51
Hypocalcemia (Metabolism and nutrition disorders) | 14 | 31
Hypokalemia (Metabolism and nutrition disorders) | 9 | 32
Hypomagnesemia (Metabolism and nutrition disorders) | 8 | 34
Hyponatremia (Metabolism and nutrition disorders) | 13 | 50
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 15
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 22 | 21
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 22 | 34
Neck pain (Musculoskeletal and connective tissue disorders) | 50 | 68
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 17 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 22
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 34 | 35
Trismus (Musculoskeletal and connective tissue disorders) | 57 | 55
Dizziness (Nervous system disorders) | 24 | 34
Dysarthria (Nervous system disorders) | 8 | 17
Dysgeusia (Nervous system disorders) | 144 | 156
Headache (Nervous system disorders) | 22 | 45
Neuralgia (Nervous system disorders) | 28 | 20
Paresthesia (Nervous system disorders) | 17 | 13
Peripheral sensory neuropathy (Nervous system disorders) | 28 | 36
Anxiety (Psychiatric disorders) | 29 | 34
Depression (Psychiatric disorders) | 30 | 36
Insomnia (Psychiatric disorders) | 23 | 46
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 46
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 24 | 37
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 36 | 36
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 45 | 42
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 27 | 29
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 53 | 50
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 14
Sore throat (Respiratory, thoracic and mediastinal disorders) | 44 | 52
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 21 | 24
Alopecia (Skin and subcutaneous tissue disorders) | 17 | 25
Dry skin (Skin and subcutaneous tissue disorders) | 13 | 37
Pruritus (Skin and subcutaneous tissue disorders) | 28 | 94
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 | 199
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 75
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 17 | 37
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 29 | 31
Skin induration (Skin and subcutaneous tissue disorders) | 59 | 65
Hypertension (Vascular disorders) | 20 | 31
Lymphedema (Vascular disorders) | 40 | 30

LIMITATIONS AND CAVEATS:
Due to a lower-than-expected death rate, the statistical design was modified to perform the primary analysis after all randomized patients had a minimum of 5 years of potential follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT00956007/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT00956007/ICF_001.pdf